CLINICAL TRIAL: NCT03904485
Title: Assessment of Myocardial Injury in Recipients of Simultaneous Pancreas and Kidney Transplantation
Brief Title: Assessment of Myocardial Injury in Simultaneous Pancreas and Kidney Transplantation
Acronym: AMI-SPK
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tianjin First Central Hospital (Other)
Responsible Party: Principal Investigator, Yingxin FU.MD, Director of kidney transplantation center, Tianjin First Central Hospital
Other Study IDs: 2019N020KY
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Simultaneous Pancreas-kidney Transplantation; Diabetic Cardiomyopathy
Keywords: SPK ,DCM,CMR
MeSH Terms: conditions — Diabetic Cardiomyopathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SPKT: patients with end-stage diabetic nephropathy got simultaneous pancreas-kidney transplantation
  Interventions: Radiation: cardiac magnetic resonance(CMR) T2 mapping
- RT: patients with end-stage diabetic nephropathy got single kidney transplantation
  Interventions: Radiation: cardiac magnetic resonance(CMR) T2 mapping

INTERVENTIONS:
Radiation: cardiac magnetic resonance(CMR) T2 mapping — T2 value before transplant，3 month and 6month after transplant

SUMMARY:
Diabetic cardiomyopathy( DCM) is a major complication of diabetes and is a common cardiovascular complication independent of coronary artery disease and hypertension．Trial to assess of myocardial injury in recipients of simultaneous pancreas and kidney transplantation by nuclear magnetic T２ mapping technology.

DETAILED DESCRIPTION:
1. Evaluate the changes of myocardial injury before and after SPK by cardiac magnetic resonance imaging (CMR),
2. Evaluate the value of SPK in the repair of myocardial injury by comparing with the single renal transplant in recipients with diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. patients with type 2 diabetes were treated with SPK; 2.No definite history of cardiovascular diseases (such as congenital heart disease, coronary heart disease, cardiomyopathy or valvular heart disease, etc.); 3. Preoperative hemodialysis 4. No history of heart failure

Exclusion Criteria:

1. Contraindications in cardiac magnetic resonance imaging；2.poorly controlled hypertension；3.CMR examination revealed marked hypertrophy of the left ventricular myocardium

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of 25 patients with SPK who met the inclusion criteria and 25 patients with simple kidney transplantation for diabetic end-stage nephropathy were included by matching the onset time, gender, age, BMI and blood pressure of diabetes
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of myocardial injury | 1year
  Assessment of myocardial injury between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin First central hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided
Study data including numbers, clinical data, and corresponding CMR results, were shared every three months

REFERENCES:
- [Background] Messroghli DR, Radjenovic A, Kozerke S, Higgins DM, Sivananthan MU, Ridgway JP. Modified Look-Locker inversion recovery (MOLLI) for high-resolution T1 mapping of the heart. Magn Reson Med. 2004 Jul;52(1):141-6. doi: 10.1002/mrm.20110. PMID 15236377
- [Background] Ding H, Fernandez-de-Manuel L, Schar M, Schuleri KH, Halperin H, He L, Zviman MM, Beinart R, Herzka DA. Three-dimensional whole-heart T2 mapping at 3T. Magn Reson Med. 2015 Sep;74(3):803-16. doi: 10.1002/mrm.25458. Epub 2014 Sep 19. PMID 25242141